CLINICAL TRIAL: NCT05207813
Title: A Prospective, Open-Label, Single-Arm Study of Intraosseous Basivertebral Nerve Ablation for the Treatment of Chronic Low Back Pain Long-term Follow Up
Brief Title: CLBP Single-Arm Long-Term Follow-up Study
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CP0015
Record Dates: First submitted 2022-01-07; First posted 2022-01-26 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Chronic Low Back Pain
Keywords: Vertebrogenic chronic low back pain; Intraosseous basivertebral nerve ablation; Low back pain; Axial low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Basivertebral nerve ablation treatment: Patient-reported outcomes at three (3) follow-up visits for previously treated participants from the CLBP Single-Arm study.
  Interventions: Device: Intracept Procedure

INTERVENTIONS:
Device: Intracept Procedure — Intraosseous Basivertebral Nerve (BVN) Ablation

SUMMARY:
This is a prospective, noninterventional, observational post market data collection of long-term effectiveness and satisfaction outcomes for "A Prospective, Open-Label, Single-Arm Study of Intraosseous Basivertebral Nerve Ablation for the Treatment of Chronic Low Back Pain (CLBP Single-Arm Study)" population at three (3), four (4), and five (5) years post Intracept Procedure. The working hypothesis is that data collected in this study will demonstrate safety, efficacy, durability and reproducibility of BVN ablation treatment outcomes out to 3, 4, and 5-years post-procedure.

DETAILED DESCRIPTION:
Patients were originally enrolled under NCT03266107 and followed through 12-months post Intracept Procedure. This study approached patients from NCT03266107 to collect additional long-term effectiveness and satisfaction outcomes at three (3), four (4), and five (5) years post Intracept Procedure.

ELIGIBILITY:
Inclusion Criteria:

- Patient received the Intracept procedure while participating in "A Prospective, Open-Label, Single-Arm Study of Intraosseous Basivertebral Nerve Ablation for the Treatment of Chronic Low Back Pain (CLBP Single-Arm Long-Term Study)"

Exclusion Criteria:

- None

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 47 subjects treated in original CLBP Single-Arm Study will be given the option to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bloom Lyons, Study Director — Boston Scientific Corporation
Locations (2):
- United States (2):
  - Indiana Spine Group, Carmel, Indiana
  - Seton Healthcare Family, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Truumees E, Macadaeg K, Pena E, Arbuckle J 2nd, Gentile J 2nd, Funk R, Singh D, Vinayek S. A prospective, open-label, single-arm, multi-center study of intraosseous basivertebral nerve ablation for the treatment of chronic low back pain. Eur Spine J. 2019 Jul;28(7):1594-1602. doi: 10.1007/s00586-019-05995-2. Epub 2019 May 21. PMID 31115683
- [Result] Macadaeg K, Truumees E, Boody B, Pena E, Arbuckle J 2nd, Gentile J, Funk R, Singh D, Vinayek S. A prospective, single arm study of intraosseous basivertebral nerve ablation for the treatment of chronic low back pain: 12-month results. N Am Spine Soc J. 2020 Sep 18;3:100030. doi: 10.1016/j.xnsj.2020.100030. eCollection 2020 Oct. PMID 35141598

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Basivertebral Nerve Ablation Treatment
Started | 42
Completed | 40
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Basivertebral Nerve Ablation Treatment
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.75 (8.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 40
Oswestry Disability Index (ODI) [Mean (Standard Deviation); unit: score on a scale] — The Oswestry Disability Index (ODI) is a validated questionnaire of pain-related disability with total score on a scale of 0 (no disability) to 100 (complete disability). Categories for ODI total score are 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). The published minimally clinically important difference for change in ODI is 10 points.
  score on a scale | 47.05 (10.17)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in ODI From Baseline to 5 Years Post Intracept Procedure
Description: The Oswestry Disability Index (ODI) is a validated questionnaire of pain-related disability with total score on a scale of 0 (no disability) to 100 (complete disability). Categories for ODI total score are 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). The published minimally clinically important difference for change in ODI is 10 points.
Time Frame: Difference between baseline and 5-year post treatment measurements. Patients originally enrolled under NCT03266107. Baseline information for this analysis is from NCT03266107. 5-years post Intracept Procedure data collected through this NCT record/study.
Population: Patients who completed all long-term follow-up visits (3-, 4-, 5-year follow-up visit).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Basivertebral Nerve Ablation Treatment
Number analyzed (Participants) | 40
units on a scale | 34.63 (10.12)

2. Secondary Outcome: Mean Change in Oswestry Disability Index (ODI) From Baseline to 3 Years Post Intracept Procedure
Description: as for outcome 1
Time Frame: Difference between baseline and 3-year post treatment measurements. Patients originally enrolled under NCT03266107. Baseline information for this analysis is from NCT03266107. 3-years post Intracept Procedure data collected through this NCT record/study.
Population: Patients who completed all long-term follow-up visits (3-, 4-, 5-year follow-up visit).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Basivertebral Nerve Ablation Treatment
Number analyzed (Participants) | 40
units on a scale | 33.25 (10.75)

3. Secondary Outcome: Mean Change in ODI From Baseline to 4 Years Post Intracept Procedure
Description: as for outcome 1
Time Frame: Difference between baseline and 4-year post treatment measurements. Patients originally enrolled under NCT03266107. Baseline information for this analysis is from NCT03266107. 4-years post Intracept Procedure data collected through this NCT record/study.
Population: Patients who completed all long-term follow-up visits (3-, 4-, 5-year follow-up visit).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Basivertebral Nerve Ablation Treatment
Number analyzed (Participants) | 40
units on a scale | 34.50 (12.26)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/assess for the subjects from the time of their last study visit in NCT03266107 through their 5 year-post Intracept treatment visit (approximately 4 years). This assessment included retrospective review, as such, duration is longer than overall CLBP Single-Arm long term follow-up study. NCT03266107 followed patients through 12-months post Intracept treatment.
Description: Definition differs from clinicaltrials.gov definitions. For this study only Serious Adverse Events (SAEs) potentially related to the procedure, device, or the spine were reported and evaluated for relatedness.
Arm/Group | Basivertebral Nerve Ablation Treatment
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A contractual agreement is in place between the PI and the Sponsor that restricts the rights to discuss or publish trial results without prior review by the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT05207813/Prot_SAP_000.pdf